CLINICAL TRIAL: NCT06401512
Title: A Guided Self-determination Follow-up Program Delivered Within a Digital Platform for People with Chronic Obstructive Pulmonary Disease in Primary Care
Brief Title: Digital Follow-up Program for People with Chronic Obstructive Pulmonary Disease in Primary Healthcare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Norway University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Beate-Christin Hope Kolltveit, Associate Professor, Western Norway University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 656382
Record Dates: First submitted 2024-04-23; First posted 2024-05-06 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: COPD Chronic Obstructive Pulmonary Disease
Keywords: COPD; Guided self-determination; Primary healthcare; Randomized controlled trial; Web-based follow-up
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Masking Description: The intervention is designed to evaluate a change in health service provision; therefore blinding of the intervention is not possible. The health care professionals, patients, and researchers were not blinded to the patients' group allocation. The statistician performing the analysis will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Guided self-determination (GSD) follow-up approach by primary care nurses.
- Control group (No Intervention): Regular follow-up by primary care physician.

INTERVENTIONS:
Behavioral: Guided self-determination (GSD) follow-up approach by primary care nurses. — The GSD counseling program consists of four scheduled consultations with a nurse and a digital platform with tools to help people better manage their health. The consultations will be facilitated by using reflection sheets to stimulate written reflection in the context of GSD.
  Arms: Intervention group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD), characterized by non-reversible airflow obstruction, contributes to high mortality and morbidity rates worldwide, including Norway. Individuals with COPD experience symptoms and complications that impede daily activities and diminish their quality of life. COPD places a growing burden on healthcare systems presently and in the future. Interventions to empower individuals to self-manage their health effectively are needed to help the challenges of living with COPD, and work towards a sustainable healthcare system. As part of the broader healthcare policy agenda, this project aligns with the increasing emphasis on digital homebased primary healthcare. The intervention in this study will combine digital homebased care and guided self-determination follow-ups (GSD) within a general practice setting.

This project consists of 1) explore the feasibility of a COPD specific GSD counselling program delivered within a digital platform in primary care, 2) explore patients' and nurses' experiences applying the program, 3) examine the treatment fidelity of the intervention amongst healthcare professionals.

This project is a pilot cluster-randomized controlled trial (RCT), including individuals diagnosed with COPD, conducted in primary healthcare settings, and assessment of feasibility and uncertainties before conducting a later full-scale cluster-RCT. The intervention draws upon the Medical Research Council's revised guidelines for developing complex intervention studies, focusing on the initial phases of intervention development and pilot testing. Primary care clinics are randomly assigned into either an intervention- or a control group. The intervention consists of the GSD counselling program with follow-up within a digital platform. The control group provide regular care. The project will include both qualitative (individual semi-structured interviews), and quantitative data (questionnaires and clinical data).

In conclusion, this project explores an innovative intervention offering personalized strategies for COPD management in primary care clinic, by containing a digitalized homebased care program and follow-ups. The study aims to improve the daily living for people with COPD, while contributing to the future sustainability of healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD living at home
* Post-bronchodilator forced expiratory volume 1 s (FEV1) to forced vital capacity (FVC) below lower limit of normality

Exclusion Criteria:

* Severe somatic disease
* Severe psychiatric diagnosis
* Not able to provide informed consent
* Do not write, speak or understand Norwegian

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Medical journal | Baseline, and 3, 6, 9 and 12 months
  COPD-related information from medical journal
Qualitative data | 6 - 18 months from baseline
  Individual interviews with participants
Questionnaire | Baseline, and 3, 6, 9 and 12 months
  Health literacy using the Health Literacy Questionnaire (HLQ).
Questionnaire | Baseline, and 3, 6, 9 and 12 months
  Impact of COPD using the COPD assessment test (CAT).
Questionnaire | Baseline, and 3, 6, 9 and 12 months
  Activity-level using International Physical Activity Questionnaire (IPAQ) - Short Form.
Questionnaire | Baseline, and 3, 6, 9 and 12 months
  Exacerbation-related information from patient
Questionnaire | Baseline, and 3, 6, 9 and 12 months
  Patient education and self-management using The Health Education Impact Questionnaire (HeiQ)
Questionnaire | Baseline, and 3, 6, 9 and 12 months
  Medication adherence using The My Experience of Taking Medicines Questionnaire (MyMEDS), adapted patients with COPD.
Questionnaire | Baseline, and 3, 6, 9 and 12 months
  Well-being using Well-Being Index (WHO-5).
Questionnaire | Baseline, and 3, 6, 9 and 12 months
  Self-rated health using EuroQol-5D-5L.
Questionnaire | Baseline, and 3, 6, 9 and 12 months
  Dyspnea using Dyspnea-12 questionnaire.
Questionnaire | Baseline, and 3, 6, 9 and 12 months
  Patient satisfaction using Client Satisfaction Questionnaire (CSQ-8) and Patient global impression of change.
Weight | Baseline and 12 months
  Weight in kg
Height | Baseline and 12 months
  Height in cm
Recruitment rate for primary care practices | Baseline
  Recruitment for primary care practices will be reported in terms of the number and proportion of primary care practices approached versus the practices that responded and, thereafter, the number who agreed to participate.
Recruitment rate for participants | Baseline
  Participant recruitment will be reported in terms of the number of participants screened, found eligible, contacted, and those who provided written consent. Data for each recruitment step will be collected from all involved practices through self-reported numbers and the signed consent forms. Proportions will also be calculated for the number of participants screened versus those contacted, as well as for those contacted versus those who provided written consent.
Retention rate | Baseline, and 3, 6, 9 and 12 months
  Retention will be reported as the number and proportion of participants who remain in the program at a certain timepoint. This will be calculated as the number of participants remaining in the program at each time point versus the number at baseline. To measure the retention rate, data from nurse reports, checklists, and medical records will be utilized.
Attrition rate | Baseline, and 3, 6, 9 and 12 months
  The attrition rate, defined as the number of participants lost to follow-up, will be calculated as 1 minus the retention rate and as the number of participants lost to follow-up between consecutive time points. To measure the attrition rate, data from nurse reports, checklists, and medical records will be utilized. Additionally, data on who exited the program at what step and from whom we lack follow-up data will be collected.
Adherence rate | Baseline, and 3, 6, and 9 months.
  Adherence rate will be collected in terms of number of sessions attended by each participant. To measure the adherence rate checklists and medical journals filled out by nurses conducting the intervention and self-reported data will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Beate-Christin H Kolltveit, Ph.D., Principal Investigator — Western Norway University of Applied Sciences
Locations (1):
- Western Norway University of Applied Sciences, Bergen, Norway, Norway

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial.
Time Frame: Data will be available two years after publication.
Access Criteria: In accordance with the approvals granted for this study by the Regional Committee on Medical Research Ethics and the Norwegian Data Inspectorate, the data files will be stored securely and in accordance with the Norwegian Law of Privacy Protection. A subset of the data file with anonymized data will be made available to interested researchers upon reasonable request to Beate-Christin Hope Kolltveit: beate-christin.hope.kolltveit@hvl.no, providing that Norwegian privacy legislation and the General Data Protection Regulation are respected, and that permission is granted from the Norwegian Data Inspectorate and the data protection officer at Western Norway University of Applied Sciences.

REFERENCES:
- [Background] Kolltveit BH, Graue M, Borge CR, Frisk B. Patients' experiences with participating in a team-based person-centred intervention for patients at risk of or diagnosed with COPD in general practice. Pilot Feasibility Stud. 2023 Sep 25;9(1):164. doi: 10.1186/s40814-023-01398-9. PMID 37749601